CLINICAL TRIAL: NCT01327755
Title: Effect of Selenium Supplementation on CD4 + Cell Recovery, Viral Suppression, Morbidity and Quality of Life of HIV Infected Patients in Rwanda: a Prospective, Double-Blinded, Placebo-Controlled Trial
Brief Title: Rwanda Selenium Supplementation Clinical Trial
Acronym: RSST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: Global Benefit Canada (Unknown); University of Ottawa (Other); Wilfrid Laurier University (Other); Kibagabaga District Hospital (Unknown); Kinyinya Health Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT-32122010
Record Dates: First submitted 2011-01-11; First posted 2011-04-04 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-02

CONDITIONS: HIV
Keywords: Selenium; HIV/ AIDS; CD4 counts; Antiretroviral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Selenium (Experimental)
  Interventions: Dietary Supplement: Selenium
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Selenium — Selenium yeast containing selenomethionine 200 mcg per day for 2 years
  Arms: Selenium
Other: Placebo — Same number of pills, frequency, and duration as selenium intervention.
  Arms: Placebo

SUMMARY:
Study Hypothesis: The addition of selenium supplementation to cotrimoxazole will improve CD4 counts, decrease opportunistic infections, decrease viral loads and delay the need for initiating antiretroviral therapy(ART) in Rwandan adult patients infected with HIV/ AIDS.

DETAILED DESCRIPTION:
Patients will be recruited from two health facilities (Kibagabaga District Hospital, and Kinyinya Health Center in Kigali), Rwanda that offer care and treatment for HIV/AIDS patients. Patients will be recruited during a 3-4 month period. Consenting adults who fit the inclusion criteria will be enrolled and followed for 2 years. Study assessments will occur at enrollment, 6, 12, 18, and 24 months after initiation of selenium supplementation.

Participants will be randomized using a simple randomized block design to receive either cotrimoxazole and selenium or cotrimoxazole and an identically appearing placebo taken once daily for 2 years. Participants who do not return to the clinic as scheduled will be followed up at home.

All consenting patients with CD4 count between 400 and 650 mm3 will be selected because they are at similar immunological level and hence they will not be eligible to start ARV treatment at the study start. The study will look at the efficacy of selenium supplementation to this already compromised group of patients at a similar stage of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = 21 years at enrollment
* Confirmed HIV positive with a CD4 range between 400 and 650 mm3
* HIV+ patients willing to participate in the study and who provide informed consent
* Pre-antiretroviral therapy (Pre-ART) at enrollment in study (not yet initiated ART)
* Willing to practice barrier method of birth control at all times

Exclusion Criteria:

* Patients intending to be transferred out of the clinic catchment area before study ends
* Patients scheduled to start ART
* Moribund patients
* Pregnant women
* Unable or not wanting to commit to barrier method of birth control

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
CD4 count | Baseline, 6, 12, 18, and 24 months

SECONDARY OUTCOMES:
viral load | Baseline, 12, and 24 months
Occurrence of opportunistic infections | Baseline, 6, 12, 18, and 24 months
Incidence of antiretroviral therapy (ART)initiation | Baseline, 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Julius K Kamwesiga, MD MPH(cand), Principal Investigator — Rwanda Selenium Supplementation Clinical Trial; Don Warren, BSc ND DHANP, Principal Investigator — Global Benefit Canada
Locations (2):
- Rwanda (2):
  - Kibagabaga Hospital, Kigali
  - Kinyinya Health Center, Kigali

REFERENCES:
- [Derived] Kamwesiga J, Mutabazi V, Kayumba J, Tayari JC, Smyth R, Fay H, Umurerwa A, Baziruwiha M, Ntizimira C, Murebwayire A, Haguma JP, Nyiransabimana J, Habarurema D, Mukarukundo V, Nzabandora JB, Nzamwita P, Mukazayire E, Mills EJ, Seely D, McCready DJ, Warren D. Effect of selenium supplementation on CD4 T-cell recovery, viral suppression, morbidity and quality of life of HIV-infected patients in Rwanda: study protocol for a randomized controlled trial. Trials. 2011 Aug 13;12:192. doi: 10.1186/1745-6215-12-192. PMID 21838913